CLINICAL TRIAL: NCT05512013
Title: The Effects of Non-steroidal Anti-inflammatory Drugs on Circulating Markers of Bone Metabolism Following Plyometric Exercise in Humans
Brief Title: The Effects of NSAIDs on Bone Metabolism Following Exercise
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jeffery Staab, Principal Investigator, United States Army Research Institute of Environmental Medicine
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 21-18H
Record Dates: First submitted 2022-08-16; First posted 2022-08-23 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Bone Resorption; Stress Fracture; Bone Injury
MeSH Terms: conditions — Bone Resorption; Fractures, Stress | interventions — Ibuprofen; Celecoxib; Flurbiprofen

STUDY DESIGN:
Intervention Model Description: 4 trial, block randomized crossover design. Three NSAIDs and one placebo trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Ibuprofen (Experimental): Participants will consume a single dose of ibuprofen prior to a plyometric exercise bout
  Interventions: Drug: Ibuprofen 800 mg
- Celecoxib (Experimental): Participants will consume a single dose of celecoxib prior to a plyometric exercise bout
  Interventions: Drug: Celecoxib 200mg
- Flurbiprofen (Experimental): Participants will consume a single dose of flurbiprofen prior to a plyometric exercise bout
  Interventions: Drug: Flurbiprofen 100 mg
- Placebo (Placebo Comparator): Participants will consume a single dose of an inert placebo prior to a plyometric exercise bout
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibuprofen 800 mg — Ibuprofen taken orally 2 hours prior to exercise
  Other Names: Advil; Motrin
  Arms: Ibuprofen
Drug: Celecoxib 200mg — Celebrex taken orally 2 hours prior to exercise
  Other Names: Celebrex
  Arms: Celecoxib
Drug: Flurbiprofen 100 mg — Flurbiprofen taken orally 2 hours prior to exercise
  Other Names: Ansaid
  Arms: Flurbiprofen
Drug: Placebo — Inert placebo taken orally 2 hours prior to exercise
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects of a single dose of non-steroidal anti-inflammatory drugs on post-exercise markers of bone and muscle metabolism.

DETAILED DESCRIPTION:
This protocol intends to determine how consuming a single dose of a non-steroidal anti-inflammatory drug (NSAID) affects circulating bone metabolism biomarkers and markers of damage skeletal muscle in response to a bout of plyometric exercise. This will be accomplished using a four trial, placebo-controlled crossover design with trials examining ibuprofen, celecoxib, flurbiprofen and placebo. These particular NSAIDs were chosen because of their widespread use in military populations and differing molecular mechanisms, which could cause differing effects on bone and muscle. Two hours after of consuming a single dose of an NSAID, participants will perform 10 sets of 10 plyometric jumps to induce a mechanical loading stimulus the bone and muscle tissues. Blood, urine, and muscle biopsy samples will be collected before and up to four hours after exercise. Biomarkers representing bone and muscle metabolism will determine the magnitude of adaptive responses to plyometric exercise while using NSAIDs.

ELIGIBILITY:
Inclusion Criteria:

* Must currently exercise at least 2 times per week
* Must be willing to discontinue the use of nutritional supplements, alcohol and nicotine during each study period (4 trials of 5 consecutive days each), unless approved by PI
* Must be willing to refrain from taking NSAIDs and similar medications during the course of the study (other than those given by the study team)
* Weigh at least 110 lbs and have a hemoglobin of 12.5 g/dL or higher

Exclusion Criteria:

* Known allergic reaction to any NSAID type medication
* History of gastrointestinal disorders/discomfort associated with or which may be aggravated with NSAID use
* History or known gastric ulcer
* History of endocrine disorders (e.g., diabetes, uncontrolled thyroid dysfunction, hypoparathyroidism, or hyperparathyroidism)
* History of bone-modifying disorder (e.g., osteogenesis imperfecta, osteoporosis, or rickets)
* Diagnosed bone fracture within last 6 months
* History of cardiovascular or renal diseases
* Pregnant or lactation in the last 6 months
* Currently taking or history of routine use of medications known to affect bone or calcium metabolism (e.g., thiazide diuretics, bisphosphonates, oral steroids)
* History of back or shoulder injury which may be aggravated by exercise
* Blood donation within 8 weeks of the study
* Current physical illness or injury limiting physical activity
* Known allergy to lidocaine

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline circulating marker of bone formation | Change from pre-exercise to 4 hours post-exercise
  Concentration (pg/mL) of serum N-terminal propeptide of type 1 collagen (P1NP)

SECONDARY OUTCOMES:
Change from baseline circulating marker of bone resorption | Change from pre-exercise to 4 hours post-exercise
  Concentration (pg/mL) of serum C-terminal propeptide of type I collagen (CTX)
Markers of muscle inflammation | Change from pre-exercise to 3 hours post-exercise
  Interlukin-6 (IL-6), Interlukin-10 (IL-10), and tissue necrosis factor (TNF-a) messenger ribonucleic acid (mRNA) concentration in muscle biopsy tissue

OTHER OUTCOMES:
Muscle protein synthesis | Change from pre-exercise to 3 hours post-exercise
  ribosomal protein S6 (p-RPS6) protein concentration in muscle biopsy tissue

CONTACTS AND LOCATIONS:
Locations (1):
- United States Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Staab JS, Kolb AL, Tomlinson RE, Pajevic PD, Matheny RW Jr, Hughes JM. Emerging evidence that adaptive bone formation inhibition by non-steroidal anti-inflammatory drugs increases stress fracture risk. Exp Biol Med (Maywood). 2021 May;246(9):1104-1111. doi: 10.1177/1535370221993098. Epub 2021 Feb 27. PMID 33641442
- [Background] Jankowski CM, Shea K, Barry DW, Linnebur SA, Wolfe P, Kittelson J, Schwartz RS, Kohrt WM. Timing of Ibuprofen Use and Musculoskeletal Adaptations to Exercise Training in Older Adults. Bone Rep. 2015 Jan 1;1:1-8. doi: 10.1016/j.bonr.2014.10.003. PMID 25642444
- [Background] Kohrt WM, Barry DW, Van Pelt RE, Jankowski CM, Wolfe P, Schwartz RS. Timing of ibuprofen use and bone mineral density adaptations to exercise training. J Bone Miner Res. 2010 Jun;25(6):1415-22. doi: 10.1002/jbmr.24. PMID 20200939
- [Background] Wherry SJ, Wolfe P, Schwartz RS, Kohrt WM, Jankowski CM. Ibuprofen taken before exercise blunts the IL-6 response in older adults but does not alter bone alkaline phosphatase or c-telopeptide. Eur J Appl Physiol. 2021 Aug;121(8):2187-2192. doi: 10.1007/s00421-021-04691-8. Epub 2021 Apr 19. PMID 33876259
- [Background] Brewer CB, Bentley JP, Day LB, Waddell DE. Resistance exercise and naproxen sodium: effects on a stable PGF2alpha metabolite and morphological adaptations of the upper body appendicular skeleton. Inflammopharmacology. 2015 Dec;23(6):319-27. doi: 10.1007/s10787-015-0248-x. Epub 2015 Aug 20. PMID 26289996
- [Background] Park J, Fertala A, Tomlinson RE. Naproxen impairs load-induced bone formation, reduces bone toughness, and diminishes woven bone formation following stress fracture in mice. Bone. 2019 Jul;124:22-32. doi: 10.1016/j.bone.2019.04.009. Epub 2019 Apr 15. PMID 30998998

DOCUMENTS (1):
  • Informed Consent Form (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/13/NCT05512013/ICF_000.pdf